CLINICAL TRIAL: NCT00863135
Title: Effect of Continuous Positive Airway Pressure (CPAP) Treatment on Blood Pressure in Patients With Sleep Apnea and Refractory Hypertension
Brief Title: Effect of CPAP on Blood Pressure in Patients With Sleep Apnea and Refractory Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Principal Investigator, Jaume Almirall, Dr., Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIS PI070219
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Obstructive Sleep Apnea; Refractory Arterial Hypertension
Keywords: obstructive sleep apnea; refractory arterial hypertension; continuous positive airways pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Positive Airway Pressure (Experimental): nocturnal continuous positive airways pressure
  Interventions: Device: CPAP
- Control (Other): Waiting list,3 months without any change in their treatment, come into the CPAP procedure after that time
  Interventions: Device: Control

INTERVENTIONS:
Device: CPAP — continuous positive airways pressure
  Arms: Continuous Positive Airway Pressure
Device: Control — Patients are 3 months without any change in their treatment, and are in the waiting list to come into the CPAP procedure after that time
  Arms: Control

SUMMARY:
The purpose of this study is to determine the effects of CPAP treatment on blood pressure in patients with sleep apnea syndrome (SAS) and refractory arterial hypertension (RAH).

Also, some of the mechanisms mediating SAS and RAH (systemic inflammation, oxidative stress, sympathetic hyperactivity) will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* refractory arterial hypertension and sleep apnea with apnea-hypopnea index over 15

Exclusion Criteria:

* excessive sleepiness
* professional drivers
* secondary arterial hypertension

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
24 hours blood pressure monitoring | basal and after three months of CPAP treatment

SECONDARY OUTCOMES:
oxidative stress and inflammatory mediators | basal and after three months of CPAP treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jaume Almirall, Dr, Principal Investigator — Corporació Parc Taulí; Juan-Carlos Martinez-Ocaña, Dr, Study Chair — Corporació Parc Tauli; Antonio Ferrer, Dr, Study Chair — Corporacio Parc Tauli
Locations (1):
- Corporacio Parc Tauli, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No